CLINICAL TRIAL: NCT03770637
Title: A Phase 2, Interventional, Randomized, Double-Blind, Placebo-Controlled Pilot Study of Glucagon RTU in Subjects Who Experience Hyperinsulinemic Hypoglycemia After Bariatric Surgery
Brief Title: Glucagon Ready to Use (RTU) in Subjects With Hyperinsulinemic Hypoglycemia After Bariatric Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: XSGR-PBH-201
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Hyperinsulinemic Hypoglycemia
Keywords: glucagon; post-bariatric hypoglycemia
MeSH Terms: conditions — Congenital Hyperinsulinism | interventions — Glucagon

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, double-blind, two-treatment, 2-period, crossover in-patient phase followed by a placebo-controlled, double-blind, parallel two-treatment outpatient stage..
Who Masked: Participant, Investigator
Masking Description: The sponsor, investigators/staff and subjects will be blinded to treatment assignment. Active study drug and placebo have the identical appearance (i.e., clear, colorless liquid), and both will be provided in identical vials with blinded labeling that does not reveal the contents of the vial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glucagon RTU (glucagon injection) (Experimental): Glucagon Ready-to-Use (RTU); 60 μL injection (0.3 mg glucagon)
  Interventions: Drug: Glucagon RTU
- Placebo (Placebo Comparator): Non-active vehicle for Glucagon RTU; 60 μL injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glucagon RTU — Glucagon RTU is a sterile subcutaneous injectable non-aqueous solution formulation supplied in a vial and administered via syringe.
  Other Names: glucagon
  Arms: Glucagon RTU (glucagon injection)
Other: Placebo — The placebo is a non-active version of Glucagon RTU formulation, containing the same solvent and excipients (i.e., vehicle).
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled Phase 2 study to assess the efficacy, safety and tolerability of Glucagon RTU when administered to subjects with a history of bariatric surgery during episodes of post-postprandial hypoglycemia. Twelve eligible subjects will be randomly assigned to receive Glucagon RTU or placebo at the first of two clinical research center (CRC) visits, followed by the other treatment at the second CRC visit. Subjects will be randomly assigned to either Glucagon RTU or Placebo for the duration of a 12-week Outpatient Stage. A follow-up safety assessment visit will occur 14 to 28 days after a subject's last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Aged 18 to 75 years of age, inclusive
3. Symptoms of hypoglycemia that developed after bariatric surgery (Roux-en-Y gastric bypass [RYGB] only) in the absence of antidiabetic medications
4. History of bariatric surgery (RYGB only), at least 6 months prior to screening
5. Whipple's triad

   1. Ability to both experience and recognize hypoglycemic awareness.
   2. Documented glucose levels < 54 mg/dL when experiencing symptoms suggestive of hypoglycemia
   3. Relief of hypoglycemia symptoms when the glucose is raised to normal
6. Diagnosis of post-bariatric hypoglycemia (PBH) by a physician, requiring intervention such as intake of oral carbohydrates. This diagnosis includes documentation of endogenous hyperinsulinism in the presence of low plasma glucose.
7. In subjects with medical history of diabetes, medical documentation of postoperative remission of diabetes mellitus (fasting glucose < 110 mg/dL), and HbA1c < 6% (or 42 mmol/mL) with all previous antidiabetic medication discontinued for at least 6 months before screening.
8. Body mass index (BMI) ≤ 40 kg/m2
9. Willingness to follow all study procedures, including attending all clinic visits and self-administering blinded study drug at home for 12 weeks
10. Understands the study procedures, alternative treatment available, and risks involved with the study, and he/she voluntarily agrees to participate by giving written informed consent
11. Women of childbearing potential must have a negative urine pregnancy test and agree to use contraception and refrain from breast-feeding during the study and for at least 15 days after participating in the study.

Exclusion Criteria:

1. Documented hypoglycemia occurring in the fasting state (> 12 hours fast) within 12 months of study entry
2. Hypoglycemic unawareness as evidenced by a Gold Scale score > 4 at screening
3. Early Dumping Syndrome
4. Known insulinoma or adrenal insufficiency
5. Active treatment with any insulin/insulin secretagogues, or other diabetes medications except for acarbose and glucagon-like peptide 1 (GLP-1) analogues
6. Chronic kidney disease Stage 4 or 5 or an estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m2 at screening
7. Hepatic disease, including serum alanine aminotransferase or aspartate aminotransferase ≥ 3 times the upper limit of normal (ULN); hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL
8. Congestive heart failure, New York Heart Association Class III or IV
9. History of myocardial infarction, unstable angina, or revascularization within 6 months prior to screening.
10. History of a cerebrovascular accident within 6 months prior to screening or with major neurological deficits
11. Seizure disorder (other than with suspected or documented hypoglycemia).
12. Active malignancy, except for basal or squamous cell skin cancers
13. Personal or family history of pheochromocytoma or disorder with increased risk of pheochromocytoma (MEN 2, neurofibromatosis, or Von Hippel-Lindau disease)
14. Major surgical operation within 30 days prior to screening
15. Hematocrit ≤ 30%
16. Bleeding disorder, treatment with warfarin, or platelet count < 50,000 /mm3
17. Active alcohol abuse or substance abuse (per investigator assessment)
18. Current chronic administration of oral or parenteral corticosteroids, however topical, intraarticular, and inhaled corticosteroids are allowed
19. Use of an investigational drug within 15 days or 5 half-lives, whichever is longer, prior to screening
20. Member of a special vulnerable populations such as pregnant women, prisoners, institutionalized or incarcerated individuals, or others who may be considered vulnerable
21. Any other medical condition or finding that in the opinion of the investigator or sponsor, would compromise the safety of the subject or compromise the integrity of the study data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Blood glucose recovery: CRC | At 15 minutes following administration of study drug
  Number of subjects with blood glucose > 70 mg/dL
Blood glucose recovery: Out-patient | At 15 minutes following administration of study drug
  Frequency of blood glucose > 70 mg/dL

SECONDARY OUTCOMES:
Symptomatic Recovery: CRC | At 15, 30, and 60 minutes following administration of study drug
  Change from Baseline in Hypoglycemia Symptoms
Incidence of severe hypoglycemia: CRC | At 0-240 minutes following administration of study drug
  Number of subjects requiring external assistance to treat hypoglycemia
Incidence of severe hypoglycemia: Out-patient | During 12 weeks of out-patient treatment
  Frequency of external assistance to treat postprandial hypoglycemia
Incidence of serious hypoglycemia: CRC | At 0-240 minutes following administration of study drug
  Number of subjects with blood glucose < 54 mg/dL
Incidence of serious hypoglycemia: Out-patient | During 12 weeks of out-patient treatment
  Frequency of postprandial blood glucose < 54 mg/dL
Hypoglycemia Fear Scale | During 12 weeks of out-patient treatment
  Change from Baseline in Hypoglycemia Fear Scale (HFS-2) Scores. The HFS-2 consists of two domains, Behavior, which has 15 questions, and Worry, which has 18 questions. Each question is assessed on a 5-point scale from 0=Never to 4=Almost Always. Lower scores indicate less fear of hypoglycemia, while higher scores indicate a greater level of fear.
EuroQol Health Questionnaire (EQ-5D) | During 12 weeks of out-patient treatment
  Change from Baseline in EQ-5D Score. This is a health assessment questionnaire with three domains. The first two domains of pain/discomfort and anxiety/depression are scored on a 5-point scale from 1=no pain/discomfort; not anxious or depressed to 5=extreme pain or discomfort; extremely anxious or depressed. For these two domains, lower scores indicate less pain/discomfort or anxiety/depression, while higher scores indicate increasing levels of pain/discomfort or anxiety/depression. The third domain of Health is assessed with a series of 5 visual analog scales, each scored from 0-100. On these VAS scales, high scores indicate better health, while low scores indicate worse health.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Colorado-Denver, Aurora, Colorado
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Mayo Clinic- Rochester, Rochester, Minnesota
  - Duke Early Phase Clinical Research, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No